CLINICAL TRIAL: NCT01313741
Title: This is a 2 Year Follow up Clinical and Radiographic Analysis of a Novel All Polyethelene Glenoid Component in Standard Total Shoulder Arthroplasty.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Knoxville Orthopedic Clinic (Other)
Responsible Party: Knoxville Orthopaedic Clinic, Knoxville Orthopaedic Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Anchor Peg Study
Record Dates: First submitted 2011-03-10; First posted 2011-03-14 (Estimated); Last update posted 2011-03-14 (Estimated); Status verified 2011-03

CONDITIONS: The Primary Disease Process Being Studied is Shoulder OA and the Effect of an All Polyethelene Glenoid Component on Shoulder Arthroplasty

ARMS (1):
- Single arm shoulder arthroplasty (Experimental)
  Interventions: Device: Shoulder arthroplasty with anchor peg glenoid

INTERVENTIONS:
Device: Shoulder arthroplasty with anchor peg glenoid — Shoulder arthroplasty with anchor peg glenoid

SUMMARY:
Two hundred patients will be analyzed both clinically (via validated outcomes measures) and radiographically (via 2 sets of standard radiographs) to determine the survival and degree of bone in growth of a novel all polyethelene glenoid component used in a standard FDA approved shoulder arthroplasty system.

DETAILED DESCRIPTION:
Methods and Materials: The standard of care in my practice and most practices is to have arthroplasty patients return for an annual clinical and radiographic evaluation. We are asking our patients that choose to enroll in the study to simply return for routine "standard of care" follow up. The only deviation from this standard of care is the method by which we obtain the xrays. In this study we will obtain true AP (anterior/posterior) and axillary views on there return visit. These are our normal "standard of care" xrays. The only difference is that we are going to obtain these Xrays using fluoroscopic guidance. The reason we are using fluoroscopic guidance is that we want to make sure that the xrays are perfect with the beam oriented tangential to the backside of the glenoid. This will allow us to see any lucencies behind the glenoid and allow us to truly assess for any loosening. Standard Xrays attempt to have the beam oriented tangential to the glenoid but just small deviations can underestimate any potential lucent lines. This will expose the study subjects to small amounts of radiation that would be outside the "standard of care". The patients will be informed of this and the dose recorded. The fluoroscopy procedure will take about 15-20 minutes, but the total radiation exposure for the activities performed will be up to, but not more than three minutes. The total radiation will be less than 3 rem. A licensed radiology technologist (RT) employed by the hospital will perform the fluoroscopy procedures and the Xrays. Jeff Jarnagin PA or Edwin Spencer MD will be present at all times during the fluoroscopy procedure. Both Dr Spencer and Jeff Jarnagin have been involved in other similar studies and have completed "training in human research subject protection". Subjects will be provided proper shielding (lead apron) throughout the activities. The licensed radiology technologist at the hospital will have the final responsibility for providing proper shielding.

As with every clinical study, there may be some risks. Since the fluoroscope emits X-rays, subjects will be exposed to radiation. During fluoroscopy, the actual dose of radiation exposure that will be administered, is within minimal risk limits and will be much lower than those known to produce detectable health effects. For this study, the fluoroscopy machine will be on for up to, but not more than, 3 minutes total and the amount of radiation will not exceed 3 rem which includes the radiation from the standard Xrays. According to published literature, exposure risks below 5-10 rem are minimal. Health effects have not been consistently demonstrated for radiation exposure below 10 rem.

Subjects will also fill out 2 data sheets. One is for the PENN score and the other is for the ASES (Association of Shoulder and Elbow Surgeons) score which are validated clinical outcomes measures. These forms are routinely filled out at their annual clinical visits and are considered standard of care.

Data Analysis: The radiographs will be independently evaluated by 2 different board certified radiologists blinded to the clinical results and names of the patients. The films will be re-evaluated by each radiologist (they will be blinded to their initial reading) and the average of their results will be recorded. The clinical ASES and PENN scores will be recorded and differences in the preoperative and postoperative scores will be reported. Statistical analysis such as a students t test is not necessary as we are not comparing two groups however simple descriptive statistics will be used to report the change in ASES and PENN scores and most importantly the presence or absence of lucent lines and location of any lucencies. The lucent lines will be graded according to the method developed by Lazarus et al.4 The medical records and Xray data will be kept as confidential as possible under current local, state, and federal laws. The researchers will examine the medical records for information related to both of the shoulders and the study data. The medical records that identify the subject and the consent form will be reviewed by the researchers. The results of this research project may be presented at meetings or in publications. The identity of the subject will not be disclosed in any presentation or publication.

The Xrays will be stored in a secure place at the Knoxville Orthopaedic Clinic. These Xrays will be accessible by only approved personnel. They will be kept indefinitely for the possibility of future use in research or publications.

Personnel who will have access to your information include:

* Jeff Jarnagin PA (Assistant to Dr Spencer)
* Dr. Edwin Spencer, PI (Orthopaedic Surgeon)

Risk Analysis: The only risk involved is the extra amount of radiation required to obtained the floroscopically guided Xrays. As stated above the maximum amount of radiation is 3 rem which includes the radiation from the standard Xrays. According to published literature, exposure risks below 5-10 rem are minimal. Health effects have not been consistently demonstrated for radiation exposure below 10 rem. To protect the subjects a licensed radiology technologist (RT) employed by the hospital will perform the fluoroscopy procedures and the Xrays. Jeff Jarnagin PA or Edwin Spencer MD will be present at all times during the fluoroscopy procedure. Subjects will be provided proper shielding (lead apron) throughout the activities. The licensed radiology technologist at the hospital will have the final responsibility for providing proper shielding.

The benefits to the patient is for the researchers (and readers of any published data) to garner a better understanding of the best method to resurface the glenoid in a TSA. Many patients require bilateral operations and therefore it could directly benefit a few patients but essentially this project is designed to gather information for the greater good of all patients who require a TSA.

Subject Identification, Recruitment And Consent: Subjects will be identified by a unique identification number analogous to that used by the Knoxville Orthopaedic Clinic. Subjects will be called by either Dr Edwin E Spencer Jr MD (PI) or his assistant Jeff Jarnagin PA and asked to be involved or participate. The patients will be made aware that participation in the study is completely voluntary and that participation does not affect their future access to care by Dr Spencer. Informed consent will be reviewed over the phone and in person when they come in for Xrays by Dr Spencer or his assistant Jeff Jarnagin PA. Attached is our consent form. Once the subject has completed the xray evaluation and completed the clinical forms, they will be paid the $50 stipend. The subject will incur no cost for participation in the study. Insurance carriers will not be billed for any part of the study. The money for the patients will come from the study sponsor DePuy Inc. The xrays including the floroscopy and radiologists' readings will be paid for by the study sponsor DePuy. The surgeon, Dr Spencer, will not be paid for his time and effort and is donating his time to science and the greater good.

ELIGIBILITY:
Inclusion Criteria: all patients with standard OA who had a shoulder arthroplasty with an anchor peg glenoid -

Exclusion Criteria:Any paient who had a concomitant rotator cuff tear, infection, revision or previous arthroplasty.

-

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-04; Primary Completion 2012-04 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
ASES Scores | Every 3 months
  Accepted validated clinical outcome measure
PENN Score | 3 months
  Accepted validated outcome measure
Radiographic integration of component | 2 weeks, 6 weeks, 3 months, 2 years
  Two sets of radiographs will be obtained to look for any signs of loosening and for bony integration of the component

CONTACTS AND LOCATIONS:
Locations (1):
- Knoxville Orthopaedic Clinic, Knoxville, Tennessee, United States

REFERENCES:
- See also: Website for our clinic — http://kocortho.com